CLINICAL TRIAL: NCT05829187
Title: Effectiveness of Momordica Charantia Extract Compared to the Standard Antimalarial Drug Combination Dihydroartemisinin Piperaquine-primaquine in Patients With Uncomplicated Falciparum Malaria, in Sumba Barat Daya District of Indonesia
Brief Title: Momordica Charantia and Dihydroartemisinin-piperaquined-primaquine for Uncomplicated Plasmodium Falciparum Malaria Patients in Southwest Sumba Regency
Acronym: MCHUPF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Syamsudin Abdillah,Ph.D, Pharm D (Other)
Collaborators: Apt. Dian Yudianto; Dr. dr Erni J. Nelwan, Sp.PD, Ph.D; Apt.Hesty Utami Ramadaniati, M.Clin, Pharm, Ph.D (Unknown)
Responsible Party: Sponsor-Investigator, Syamsudin Abdillah,Ph.D, Pharm D, Prof. Apt. Syamsudin, M.Biomed, Ph.D, Pancasila University
Organization: Pancasila University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B-056/FI2/KEPK/TL.00/10/2022
Record Dates: First submitted 2023-01-09; First posted 2023-04-25 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Uncomplicated Plasmodium Falciparum
Keywords: Parasite number, clinical symtomps, immunomodulator
MeSH Terms: interventions — artenimol; piperaquine; Primaquine; bitter melon extract

STUDY DESIGN:
Intervention Model Description: the patient comes to the primary health care facility, is examined by a doctor, if malaria is suspected, a parasite examination is carried out in the laboratory. If positive for falciparum malaria and based on the results of the doctor's examination meet the criteria as research subjects, then the drug is given based on the random table that has been provided.
Who Masked: Participant
Masking Description: The test drug and the control drug are put into the capsule with the same weight, type and smell so that the patient cannot distinguish between the test drug and the control drug
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dihydro artemisinin Piperakuin (Fixed Dose Combination) and Primaquine (Experimental): Fixed Dose Combination content in the form of 40 mg dihydroartemisinin and 320 mg piperaquine administered for 3 days with a dose of dihydroartemisinin 2-4 mg/Kg body weight, piperaquine at a dose of 16-32 mg/Kg body weight in the form of a combination set out in the table based on body weight and age. Primaquine dose of 0.25 mg/Kg body weight is given only on the first day. Dihydroartemisinin-piperaquine was local product by PT Mersi Pharmaceuticals, batch No 220610, produced on Jun/22 and expiring on Jun/24. primaquine was local product by PT Phapros Indonesia, Batch No 56386001, produced on Jan/22 and expiring date jan/25.
  Interventions: Drug: Dihydroartemisinin; Drug: Piperaquine; Drug: Primaquine
- Extract Capsul Momordica Charantia (Experimental): Momordica Charantia 325 mg in 500 mg capsules is given to patients with uncomplicated plasmodium falsiparum malaria as one capsule per day for three days for body weight less than 60 kg. Patients with a body weight of more than 60 kg are given two capsules per day for three days.
  Interventions: Drug: Momordica Charantia Extract

INTERVENTIONS:
Drug: Dihydroartemisinin — dihidroartemisinin dose of 2-4 mg/Kg Body weight taken for 3 days
  Other Names: 1st group
  Arms: Dihydro artemisinin Piperakuin (Fixed Dose Combination) and Primaquine
Drug: Piperaquine — piperaquine at a dose of 16-32 mg/Kg body weight taken for 3 days
  Other Names: 1st group
  Arms: Dihydro artemisinin Piperakuin (Fixed Dose Combination) and Primaquine
Drug: Primaquine — Primaquine dose 0.25 mg/kg body weight given to uncomplicated Plasmodium falciparum patients on the first day only
  Other Names: 1st Group
  Arms: Dihydro artemisinin Piperakuin (Fixed Dose Combination) and Primaquine
Drug: Momordica Charantia Extract — Momordica charantia extract capsules at a dose of 325 mg were given to patients for 3 days
  Other Names: 2nd group
  Arms: Extract Capsul Momordica Charantia

SUMMARY:
Currently, the first-line combination of artemisinin, piperaquine and prima-quine is quite effective in controlling malaria, however, the threat of spread of drug-resistant parasites has been reported. A study is conducted to assess the efficacy and safety extract of bitter melon (Momordica charantia/MC) regimens compared to the combination of dihydroartemisinin piperaquine primaquine (DHP+PQ) on the sexual and asexual stage of P. Falciparum uncomplicated in Sumba Barat Daya District, Indonesia

DETAILED DESCRIPTION:
The Study was conducted in Kori Primary Health Cender, Sumba Barat Daya District, East Nusa Tenggara Province on Sumba Island.

The study subject received either 3 day of dihydroartemisinin-piperaquine and primaquine 1 day on first day (DHP+PQ) or extract of bitter melon (Momordica charantia/MC) + Placebo 1 day on first day according to their body weight.

Patients with fever or history of fever within the past 24 hours were screened by microscopic examination of giemsa stained tihick blood films to detect Plasmodium falciparum infection.

All Patient were allocated by single blind randomization to receive DHP (on day 0 to day 2)+PQ (on day 0 only) or extract of bitter melon (Momordica charantia/MC) (on day 0 to day 2)+placebo (on day 0 only). The procedures of drug administration in the study were as follows:

ELIGIBILITY:
Inclusion Criteria:-

1. Age ≥ 18 years old male or female up to 60 years old
2. Single Plasmodium falciparum infection based on microscopic examination.
3. Count the parasites for Plasmodium falciparum at least 2 large visual field asexual parasites (LPB) by examining 15 LPB
4. Density of parasites 1000-100,000/micro liter
5. Has no history of uncontrolled comorbidities
6. History of fever in the last 24 hours for falciparum malaria
7. Not taking other antimalarial drugs in the last 2 weeks.
8. Have no previous history of malaria.
9. Willing to come to the health facility according to the specified follow-up schedule.
10. Willing to participate in research and established procedures.
11. There is no history of allergy to antimalarial drugs.

Exclusion Criteria:

1. Signs of general weakness, or decreased consciousness or recurrent seizures or circulation failure or pulmonary edema or signs of anemia or yellow body and slightly red urine.
2. If the examination results show mixed Plasmodium and non-Plasmodium falciparum.
3. Has a history of severe liver, kidney and heart dysfunction, bradycardia and heart rhythm disturbances.
4. Does not control regularly according to the research schedule
5. Pregnant and lactating women
6. There are signs of severe malaria
7. Patients with chronic diseases, for example: heart, kidney, liver, HIV.
8. Mixed infection.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
development of sexual and asexual stages of Plasmodium falciparum | 28 day post treatment
  Finger prick blood samples are collected for malaria blood smear. Thick and thin blood smear were stained with 3% giemsa solution for 45 minutes and were read under binocular microscope with 1,000x magnification

SECONDARY OUTCOMES:
Parasite clearence times | 28-days
  parasite reduction ratio
Fever clearence time | 28 days
  time taken for the axilla temperature to fall below 37.5°C in patients who were febrile at inclusion
Number of adverse event | 28 days

OTHER OUTCOMES:
Measure imunomodulator Effect | 1x24 hour before and after treatment
  Measuring the immunomodulatory effect by measuring the levels of TNF alpha and interferon gamma cytokines before and after the treatment intervention 1 x 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Kori Puskesmas, Tambolaka, East Nusa Tenggara, Indonesia

REFERENCES:
- [Background] Abdillah S, Tambunan RM, Sinaga YM, Farida Y. Ethno-botanical survey of plants used in the traditional treatment of malaria in Sei Kepayang, Asahan of North Sumatera. Asian Pac J Trop Med. 2014 Sep;7S1:S104-7. doi: 10.1016/S1995-7645(14)60213-3. PMID 25312101
- [Background] Sutanto I, Suprijanto S, Kosasih A, Dahlan MS, Syafruddin D, Kusriastuti R, Hawley WA, Lobo NF, Ter Kuile FO. The effect of primaquine on gametocyte development and clearance in the treatment of uncomplicated falciparum malaria with dihydroartemisinin-piperaquine in South sumatra, Western indonesia: an open-label, randomized, controlled trial. Clin Infect Dis. 2013 Mar;56(5):685-93. doi: 10.1093/cid/cis959. Epub 2012 Nov 21. PMID 23175563
- [Background] Jia S, Shen M, Zhang F, Xie J. Recent Advances in Momordica charantia: Functional Components and Biological Activities. Int J Mol Sci. 2017 Nov 28;18(12):2555. doi: 10.3390/ijms18122555. PMID 29182587
- [Background] Chen F, Huang G, Yang Z, Hou Y. Antioxidant activity of Momordica charantia polysaccharide and its derivatives. Int J Biol Macromol. 2019 Oct 1;138:673-680. doi: 10.1016/j.ijbiomac.2019.07.129. Epub 2019 Jul 22. PMID 31344411
- [Background] Wang S, Liu Q, Zeng T, Zhan J, Zhao H, Ho CT, Xiao Y, Li S. Immunomodulatory effects and associated mechanisms of Momordica charantia and its phytochemicals. Food Funct. 2022 Nov 28;13(23):11986-11998. doi: 10.1039/d2fo02096c. PMID 36350105
- [Result] Nelwan EJ, Ekawati LL, Tjahjono B, Setiabudy R, Sutanto I, Chand K, Ekasari T, Djoko D, Basri H, Taylor WR, Duparc S, Subekti D, Elyazar I, Noviyanti R, Sudoyo H, Baird JK. Randomized trial of primaquine hypnozoitocidal efficacy when administered with artemisinin-combined blood schizontocides for radical cure of Plasmodium vivax in Indonesia. BMC Med. 2015 Dec 11;13:294. doi: 10.1186/s12916-015-0535-9. PMID 26654101